CLINICAL TRIAL: NCT04158635
Title: A Phase 1 Study of Gemcitabine, Nab-Paclitaxel, and Bosentan in Patients With Unresectable Pancreatic Cancer
Brief Title: Gemcitabine, Nab-Paclitaxel, and Bosentan for the Treatment of Unresectable Pancreatic Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21314; NCI-2021-06609 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 19312 (Other: City of Hope Medical Center)
Record Dates: First submitted 2019-11-07; First posted 2019-11-12 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Stage III Pancreatic Cancer AJCC v8; Stage IV Pancreatic Cancer AJCC v8; Unresectable Pancreatic Carcinoma
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Bosentan; Gemcitabine; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Treatment (bosentan, nab-paclitaxel, gemcitabine) - Participant 1-9 (Experimental): Patients receive bosentan PO BID on days 8-21 of cycle 1 and days 1-21 of subsequent cycles.
  Patients also receive nab-paclitaxel IV over 30 minutes and gemcitabine IV over 30 minutes on days 1, 8, and 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Bosentan; Drug: Gemcitabine; Drug: Nab-paclitaxel; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Treatment (bosentan, nab-paclitaxel, gemcitabine) - Participant 10-12 (Experimental): Patients receive bosentan PO BID on days -7 to 21 and days 1-21 of subsequent cycles.
  Patients also receive nab-paclitaxel IV over 30 minutes and gemcitabine IV over 30 minutes on days 1, 8, and 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Bosentan; Drug: Gemcitabine; Drug: Nab-paclitaxel; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Treatment (bosentan, nab-paclitaxel, gemcitabine) - Participant 13-21 (Experimental): Patients receive bosentan PO BID on days 1-21 of cycle 1 and days 1-21 of subsequent cycles.
  Patients also receive nab-paclitaxel IV over 30 minutes and gemcitabine IV over 30 minutes on days 1, 8, and 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Bosentan; Drug: Gemcitabine; Drug: Nab-paclitaxel; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Bosentan — Given PO
  Other Names: Bosentan Monohydrate; Ro 47-0203; Tracleer
Drug: Gemcitabine — Given IV
  Other Names: dFdC; dFdCyd; Difluorodeoxycytidine
Drug: Nab-paclitaxel — Given IV
  Other Names: ABI 007; ABI-007; Abraxane; Albumin-bound Paclitaxel; Albumin-Stabilized Nanoparticle Paclitaxel; Nanoparticle Albumin-bound Paclitaxel; Nanoparticle Paclitaxel; Paclitaxel Albumin; paclitaxel albumin-stabilized nanoparticle formulation; protein-bound paclitaxel
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase I trial studies the side effects and best dose of bosentan and how well it works when given together with gemcitabine and nab-paclitaxel for the treatment of pancreatic cancer that cannot be removed by surgery (unresectable). Bosentan may block the hormone endothelin and prevent the growth and spread of pancreatic cancer. Drugs used in chemotherapy, such as gemcitabine and nab-paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving bosentan with chemotherapy (gemcitabine and nab-paclitaxel) may work better in treating patients with pancreatic cancer compared to chemotherapy alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the safety, toxicity and feasibility of administering bosentan with nab-paclitaxel and gemcitabine.

SECONDARY OBJECTIVES:

I. To assess the response rate associated with this combination therapy in first line pancreatic cancer patients.

II. To assess the progression-free survival and overall survival of all patients who start protocol therapy, and describe the outcomes based on measures of compliance during the lead-in week, and compliance with supplement during chemotherapy.

EXPLORATORY OBJECTIVES:

I. To determine the impact of bosentan on the mass transport in the tumor (surrogate of alterations in tumor stroma and blood flow). (Pharmacodynamic Investigations) II. To describe the pharmacokinetic profile of nab-paclitaxel and bosentan and compare to historic single-agent profile. (Pharmacokinetic Investigations) III. To explore the association between hepatotoxicity to study agents and organic anion-transporting polypeptide (OATP) polymorphisms. (Pharmacogenomic Investigations) IV. To explore biomarkers on pre-treatment biopsy samples and peripheral blood samples for correlations of predictive of response.

V. To describe quality of life utilizing the Functional Assessment of Cancer Therapy: General (FACT-G) questionnaire.

OUTLINE:

Patients receive bosentan orally (PO) twice daily (BID) on days -7 to 21 or 8-21 of cycle 1 and days 1-21 of subsequent cycles. Patients also receive nab-paclitaxel intravenously (IV) over 30 minutes and gemcitabine IV over 30 minutes on days 1, 8, and 15. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days. Patients who complete study treatment without disease progression are followed up every 2 months until disease progression and then biannually thereafter. Patients who complete study treatment with disease progression are followed up biannually.

ELIGIBILITY:
Main Inclusion Criteria

* Adult patients with unresectable pancreatic carcinoma
* Patients must be a candidate to receive one of the following chemotherapy combinations as determined by the treating physician:

Arm A2: gemcitabine plus nab-paclitaxel given every 2 weeks (arm A1 is closed per this amendment)

Arm B: mFOLFIRINOX given every 2 weeks

* Willingness to permit study team to obtain and use archival tissue, if already existing, or, be willing to undergo a fresh tumor biopsy if clinically possible (exceptions may be provided by study PI if medically unsafe to perform biopsy).
* Weight ≥ 40 kg
* ANC ≥ 1500/mm3; platelets ≥ 100,000/mm3
* AST, ALT ≤ 1.5 x ULN. Patients with liver metastases ≤ 3 x ULN
* Total serum bilirubin ≤ 1.5 x ULN
* Creatinine clearence ≥ 60 mL/min

Main Exclusion Criteria

* Current or planned use of Warfarin, Cyclosporine A, Rifampicin, Glyburide (other diabetic medications are allowed)
* Current or planned use of agents contraindicated for use with strong CYP3A4 inducers
* Strong inhibitors or inducers of CYP2C9
* Strong inhibitors or inducers of CYP3A
* Agent or agents that moderately inhibit both CYP2C9 and CYP3A (via a single concomitant agent, or co-administration of concomitant agents)
* No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated Stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease free for five years.
* Current or history of ≥ Grade 2 peripheral neuropathy
* Known allergy to eggs or any of the components within the study agents and/or their excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2026-01-27 (Estimated); Study Completion 2026-01-27 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 30 days after last dose of protocol therapy
  Will be recorded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v) 4.0.
Dose limiting toxicities (DLTs) | Up to 21 days (Cycle 1)
  Toxicities will be graded according to NCI CTCAE v 4.0. DLT's apply only to bosentan-only single stage AND cycle 1 and should be attributable to the treatment.
Compliance | During the first week
  Number of bosentan tablets and bottles returned will be reconciled with the patient diary.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Time to disease progression/ relapse or death as a result of any cause, assessed up to 2 years
  Will be evaluated using the Kaplan-Meier methods, both as a single group and by disease classification (metastatic versus [vs.] advanced unresectable). Response will also be examined by disease classification as part of a secondary analysis.
Overall survival (OS) | Time to death as a result of any cause, assessed up to 2 years
  Will be evaluated using the Kaplan-Meier methods, both as a single group and by disease classification (metastatic vs. advanced unresectable). Response will also be examined by disease classification as part of a secondary analysis.
Time to treatment failure (TTF) | Time to treatment termination for any reason (progression, toxicity, death, patient preference), assessed up to 2 years
  Will be evaluated using the Kaplan-Meier methods, both as a single group and by disease classification (metastatic vs. advanced unresectable). Response will also be examined by disease classification as part of a secondary analysis.

OTHER OUTCOMES:
Temporal impact of bosentan therapy on tumor vs. normal pancreatic tissue perfusion profile (tumor stroma and blood flow) | Up to 2 years
Levels of nab-paclitaxel, bosentan and active plasma metabolite Ro 48-5033 | Up to 2 years
  Will be quantitated in the peripheral blood.
Analysis of loci that encode organic anion transporting polypeptides (OATP) in participants who experience severe hepatotoxicity, increased during protocol therapy | Up to 2 years
Quantification of the number of circulating tumor cells and temporal proteomic/micro ribonucleic acid (miRNA) profile will assess response to therapy | Up to 2 years
Histopathology/ structural assessment and quantification of the miRNA profile | Up to 2 years
  Will allow the identification of prognostic biomarkers.
Quality of life assessment | Up to 2 years
  Assesses using Functional Assessment of Cancer Therapy: General (FACT-G) questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Salgia, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States